CLINICAL TRIAL: NCT00888862
Title: Desvenlafaxine Succinate in Major Depressive Disorder: Effects on Structural and Functional Imaging, Cognition, and Functional Outcomes in Midlife Women and Men
Brief Title: Desvenlafaxine Succinate (DVS) for Major Depressive Disorder (MDD) in Midlife Men and Women
Acronym: DVS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); St. Joseph's Healthcare Hamilton (Other); McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHCC2008-3
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2009-04

CONDITIONS: Major Depressive Disorder; Menopausal Staging and Vasomotor Symptoms (for Females)
Keywords: depression; desvenlafaxine; menopause; imaging; FMRI
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Use of desvenlafaxine succinate, flexible dose (50-100mg/day)
  Interventions: Drug: Desvenlafaxine Succinate

INTERVENTIONS:
Drug: Desvenlafaxine Succinate — Desvenlafaxine Succinate, 50-100mg/day for 8 weeks
  Other Names: Pristiq

SUMMARY:
The main objective of this study is to characterize a range of brain activation symptoms associated with depression and response to treatment in midlife men and women with MDD, using MRI and functional MRI. Moreover, in the female sub-group, the investigators will examine whether these brain activation symptoms are related to menopausal symptoms (i.e., hot flashes and night sweats). Also, assessing brain activation before and after the treatment might help to uncover some mechanisms associated with the pathophysiology of depression and menopause.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) has been associated with morphological changes in the brain and changes in key brain areas. Studies have shown that antidepressant use may promote the normalization of these areas. Moreover, midlife men and women appear to be at greater risk for developing major depressive episodes. In women, this period of life has been associated with significant functional impairment due to the presence/severity of vasomotor symptoms (hot flashes, night sweats), cognitive complaints, and poorer quality of life. Desvenlafaxine succinate (DVS) has been developed for the treatment of MDD. To date, the effects of DVS on brain structure and functioning in midlife men and women with MDD, as well as on depression related to menopause, has not been explored. The present study aims to investigate the effects of DVS on brain structure and functioning when used for the treatment of a major depressive episode in midlife men and women, using MRI and functional MRI. In addition, the investigators will examine whether the impact of treatment with DVS on vasomotor symptoms, cognition, and quality of life modulate the putative changes in brain structure and functioning.

ELIGIBILITY:
Inclusion Criteria:

* men and women, aged 40-60 years
* diagnosis of MDD
* for women, perimenopausal or postmenopausal

Exclusion Criteria:

* other DSM-IV axis I diagnosis other than MDD
* using psychotropic medications
* suicidal ideation, homicidal ideation, or psychotic symptoms
* presence of laboratory abnormalities at baseline visit
* presence of heart disease, liver disease, kidney disease, pulmonary disease, blood or bleeding disease, thyroid disease, GI disease, seizure or epilepsy, head injury, cancer, uterine fibroids or endometriosis, gynecologic surgeries (except caesarian sections), electroconvulsive therapies in the past 3 months, HIV+/AIDS
* in addition (for women): use of hormone replacement therapies, menstrual dysfunction, pregnancy or breastfeeding

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Effects of desvenlafaxine succinate (DVS) on brain structure and activation in midlife men and women with MDD. | 10 weeks

SECONDARY OUTCOMES:
Changes in brain activity | 10 weeks
Changes in menopause-related symptoms among females | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claudio N Soares, MD, PhD, Principal Investigator — St. Joseph's Healtcare; McMaster University
Locations (1):
- Women's Health Concerns Clinic, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Frey BN, Hall GB, Attard S, Yucel K, Skelin I, Steiner M, Soares CN. Shift in the brain network of emotional regulation in midlife women: is the menopausal transition the turning point? Menopause. 2010 Jul;17(4):840-5. doi: 10.1097/gme.0b013e3181df840f. PMID 20616670